CLINICAL TRIAL: NCT04607577
Title: Cross-cultural Adaptation and Validation in Moroccan Arabic Dialect "Darija" of the QoR-15 Postoperative Recovery Quality Score"
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Moroccan Society of Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: QoR-15MA
Record Dates: First submitted 2020-10-20; First posted 2020-10-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Recovery of Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The QoR-15 Is a post operative recovery score developed in 2013 from the QoR-40 with an advantage of simplification. The investigators Aim to translate and to validate a such useful score in Arabic adapted for Morocco by a full psychometric evaluation of the Arabic version, by testing its validity, reliability, responsiveness, and clinical acceptability and feasibility, with patients undergoing abdominal, thoracic, gynecological surgery, or digestive endoscopy in the National Institute of Oncology of Rabat, affiliated to Mohammed V University in Rabat, Morocco.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Agreement in writing for the use of the data

Exclusion Criteria:

* Patients who expressed their refusal to participate in the study
* Patients unable to express their non-opposition to participating in the study
* Patients operated on for surgery for which it was highly probable that it would not be possible for them to answer the questionnaire postoperatively (first 24 hours)
* Patients who do not master the Arabic language, neither read nor spoken

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All scheduled anesthesia procedures with a pre-anesthetic consultation, performed at INO, both in the digestive surgery operating room, as well as in gyneco-mammary and outpatient endoscopy, brachytherapy and conventional and interventional adult radiology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-01-22 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Quality of Recovery 15 in Moroccan Arabic scale (QoR-15 MA) functional recovery score at recovery from anesthesia | One Hour after recovery from anesthesia
The differential between the QoR-15MA score preoperatively and postoperatively | Day 1
  Change from preoperative baseline of QoR-15MA to postoperative scale at one hour after recovery from anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Abdelilah Ghannam, MD, Principal Investigator — Mohammed V University in Rabat
Locations (1):
- National Institute of Oncology of Rabat, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided